CLINICAL TRIAL: NCT04429568
Title: Cardiovascular Effects of Cannabis Compared to Tobacco Use
Brief Title: THC Crossover Study
Acronym: TRDRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17-24117
Record Dates: First submitted 2019-08-20; First posted 2020-06-12 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: THC; Cannabis; Cannabis Smoking; Cannabis Use, Unspecified; Cigarette Smoking; Tobacco Use; Nicotine Dependence; Nicotine Withdrawal; Cardiovascular Risk Factor
Keywords: vape; cannabis; tobacco cigarette; thc; marijuana; smoking
MeSH Terms: conditions — Marijuana Abuse; Marijuana Smoking; Cigarette Smoking; Tobacco Use; Tobacco Use Disorder; Vaping; Wiskott-Aldrich Syndrome; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smoked Cannabis, Vaped Cannabis, or Tobacco Cigarette (Other): * Abstinence from any product night before hospital admission
  * Standardized Session of assigned product: smoked cannabis, vaped cannabis, or tobacco cigarette
  * 6-hr abstinence and blood draws (PK)
  * 2 hr Free use session w/ video monitoring
  * Free use of assigned product
  * 12-hr cardiovascular (CV) monitoring
  * Circadian blood draws
  * 12-hr urine collection
  Interventions: Other: Smoked Cannabis; Other: Vaped Cannabis; Other: Tobacco Cigarette
- Either of the 2 remaining products (Other): * Abstinence from any product night before hospital admission
  * Standardized Session of assigned product: smoked cannabis, vaped cannabis, or tobacco cigarette
  * 6-hr abstinence and blood draws (PK)
  * 2 hr Free use session w/ video monitoring
  * Free use of assigned product
  * 12-hr CV monitoring
  * Circadian blood draws
  * 12-hr urine collection
  Interventions: Other: Smoked Cannabis; Other: Vaped Cannabis; Other: Tobacco Cigarette
- Remaining product (Other): * Abstinence from any product night before hospital admission
  * Standardized Session of assigned product: smoked cannabis, vaped cannabis, or tobacco cigarette
  * 6-hr abstinence and blood draws (PK)
  * 2 hr Free use session w/ video monitoring
  * Free use of assigned product
  * 12-hr CV monitoring
  * Circadian blood draws
  * 12-hr urine collection
  Interventions: Other: Smoked Cannabis; Other: Vaped Cannabis; Other: Tobacco Cigarette

INTERVENTIONS:
Other: Smoked Cannabis — Cannabis will be purchased by the participants and reimbursed the full cost by the study. Participants will be asked to purchase enough to last 2 full days of use. To reduce variability between products, participants will be asked to purchase cannabis from one dispensary near the research facility (Purple Star MD at 2520 Mission St., San Francisco). Receipt must be provided to study staff.
Other: Vaped Cannabis — Cannabis will be purchased by the participants and reimbursed the full cost by the study. Participants will be asked to purchase enough to last 2 full days of use. To reduce variability between products, participants will be asked to purchase cannabis from one dispensary near the research facility (Purple Star MD at 2520 Mission St., San Francisco). Receipt must be provided to study staff. All participants will use the study-provided PAX® (PAX 2) dry herb vaporizer, one of the most popular handheld vaporizers.
Other: Tobacco Cigarette — Tobacco cigarettes of participants' choice (usual brand) will be provided by research staff for use on the study.

SUMMARY:
This is a randomized, crossover study enrolling experienced dual cannabis-tobacco smokers (N=18) to describe the differences in THC and toxicant exposure, examining pharmacokinetic, subjective, and cardiovascular effects from smoking and vaping dry herb cannabis. This study will also examine the differences in toxicant exposure and cardiovascular disease risk between smoking cannabis and smoking tobacco cigarettes.

DETAILED DESCRIPTION:
Experienced dual cannabis-tobacco smokers will participate in a within-subject crossover study with three blocks: smoked cannabis (purchased by participants from a local dispensary), dry herb cannabis vaporizer, and usual brand tobacco cigarette. Each block will consist of 2 consecutive days on an inpatient research ward. The first inpatient day of each block will comprise of two sessions: (1) The first session will be a standardized bout to compare pharmacokinetic, physiologic, and subjective effects of cannabis and tobacco use; (2) after 6 hours of abstinence, the second session will be ad libitum access to the assigned product for 2 hours to compare subjective effects (reward, satisfaction, craving reduction) and use patterns. The second inpatient day will consist of ad libitum use of the assigned product from 8:00 in the morning to midnight. An abstinence day will be added after the second day of the last block to assess exposure and effects biomarkers during a period of abstinence from cannabis (smoked/vaped) or tobacco.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history and limited physical examination, as described below:

Heart rate < 105 beats per minute (BPM); Systolic Blood Pressure < 160 and > 90*; Diastolic Blood Pressure < 100 and > 50*

*Considered out of range if both machine and manual readings are above/below these thresholds.

* Current regular user of cannabis who smokes cannabis as joint or blunt at least 3 times a week for past 3 months
* History of cannabis vaporizer use or willingness to use the vaporizer in the study
* Current tobacco cigarette use who smokes ≥ 5 cigarettes per day
* Saliva cotinine ≥ 50 ng/ml
* Test positive for D-9-tetrahydrocannabinol (THC) at screening and self-report of cannabis use

Exclusion Criteria:

* Unstable medical conditions:

Heart disease; Uncontrolled hypertension; Thyroid disease (okay if controlled with medication); Diabetes; Hepatitis B or C or Liver disease; Glaucoma; Prostatic hypertrophy

* Psychiatric conditions:

Current or past schizophrenia, and/or current or past bipolar disorder; Adult onset attention deficit hyperactivity disorder (ADHD); Participants with current or past depression and/or anxiety disorders will be reviewed by the study physician and considered for inclusion; History of psychiatric hospitalizations are not exclusionary, but study participation will be determined as per study physician's approval

* Concurrent regular use of smokeless tobacco or pipes [occasional users of these products may be enrolled if they agree to abstain from their use during the period of the study]
* Medications:

Use of medications that are inducers of nicotine metabolizing enzyme CYP2A6 (Example: rifampicin, dexamethasone, phenobarbital, and other anticonvulsant drugs).; Concurrent use of nicotine-containing medications; Psychiatric medications: current regular use of any psychiatric medications with the exception of Selective Serotonin Reuptake Inhibitors (SSRI) and serotonin-norepinephrine reuptake inhibitors (SNRI) and current evaluation by the study physician that the participant is otherwise healthy, stable, and able to participate.

* Other/Misc. Chronic Health Conditions:

Oral thrush; Fainting; Untreated thyroid disease; Other "life threatening illnesses" as per study physician's discretion

* Pregnancy:

Pregnancy (self-reported and urine pregnancy test); Breastfeeding (determined by self-report)

* Drug/Alcohol Dependence:

Alcohol or illicit drug dependence within the past 12 months with the exception of those who have recently completed an alcohol/drug treatment program; Positive toxicology test at the screening visit (THC & prescribed medications okay); Methadone replacement therapy

* Concurrent participation in another clinical trial
* Inability to communicate in English
* History of marijuana-induced psychosis or paranoia after smoking marijuana
* Scoring a 2 or higher on the Severity of Dependence Scale for cannabis use
* Planning to quit smoking or vaping within the next 60 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration | Day 1 of each arm
  To assess the differences between smoked and vaped cannabis, we will determine maximum plasma THC concentration (Cmax) using plasma THC concentrations from the standardized sessions.
Time to peak plasma concentration | Day 1 of each arm
  To assess the differences of these variables between smoked and vaped cannabis, we will determine the time to max concentration (Tmax) using plasma THC concentrations from the standardized sessions.
Area under the plasma concentration versus time curve (AUC) | Day 1 of each arm
  To assess the differences of these variables between smoked and vaped cannabis, we will determine the AUC using plasma THC concentrations from the standardized sessions.
Subjective effects between cannabis products using the Marijuana Cravings Questionnaire | Days 1-2 of each arm
  We will assess measures from the Marijuana Cravings Questionnaire (MCQ) and compare them between smoked and vaped cannabis.
Subjective effects between cannabis products using the Visual Analog Scale | Days 1-2 of each arm
  We will assess measures from the Visual Analog Scale (VAS) and compare them between smoked and vaped cannabis.
Subjective effects between cannabis products using the Drug Effects Questionnaire | Days 1-2 of each arm
  We will assess measures from the Drug Effects Questionnaire (DEQ) and compare them between smoked and vaped cannabis.
Max change of expired carbon monoxide | Days 1-2 of the cannabis arms
  We will examine differences in max change of expired carbon monoxide (CO) from day 1 between smoked and vaped cannabis.
Area under the expired carbon monoxide (CO) curve (AUC) | Days 1-2 of the cannabis arms
  We will examine differences in integrated AUC of expired carbon monoxide from day 1 between smoked and vaped cannabis.
Differences in metabolites of volatile organic compounds (VOCs) | Days 1-2 of the cannabis arms
  We will examine differences in 12-hour urine mercapturic acid metabolites of volatile organic compounds (from day 2) between smoked and vaped cannabis.
Exposure to toxicants between cannabis products | Days 1-2 of the cannabis arms
  We will also examine how measures of use (number of puss, amount use, number of use episodes) correlate with biomarker concentrations between smoked and vaped cannabis.
Cardiovascular effects between cannabis products using heart rate as a measure | Day 1 of each arm
  We will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 30 minutes after the standardized session (day 1) between smoked and vaped cannabis.
Cardiovascular effects between cannabis products using epinephrine as a measure | Day 2 of each cannabis arm
  Urine catecholamine excretion, particularly epinephrine, will be examined in 12-hour urines and compared between smoked and vaped cannabis.
Cardiovascular effects between cannabis products using platelet activation as a measure | Day 2 of each cannabis arm
  We will examine differences in blood and urine biomarkers of platelet activation between smoked and vaped cannabis.
Cardiovascular effects between cannabis products using oxidant stress as a measure | Day 2 of each cannabis arm
  We will examine differences in blood and urine biomarkers of oxidant stress between smoked and vaped cannabis.
Cardiovascular effects between cannabis products using endothelial dysfunction as a measure | Day 2 of each cannabis arm
  We will examine differences in blood and urine biomarkers of endothelial dysfunction and inflammation between smoked and vaped cannabis.

SECONDARY OUTCOMES:
Toxicant exposure between smoked tobacco and cannabis using expired carbon monoxide as the measure | Day 1 of each arm
  We will examine differences in expired carbon monoxide (CO) from day 1 (both max change and integrated AUC of expired CO) between smoked tobacco and cannabis.
Toxicant exposure between smoked tobacco and cannabis using mercapturic acid as the measure | Day 2 of each arm
  We will examine differences in 12-hour urine mercapturic acid metabolites of volatile organic compounds (VOCs) (from day 2) between smoked tobacco and cannabis.
Toxicant exposure between smoked tobacco and cannabis using use as a measure | Days 1-2 of each arm
  We will also examine how measures of use (number of puffs, amount use, number of use episodes) correlate with biomarker concentrations between smoked tobacco and cannabis.
Cardiovascular effects between smoked tobacco and cannabis using heart rate as a measure | Day 1 of each arm
  We will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 30 minutes after the standardized session (day 1) between smoked tobacco and cannabis.
Cardiovascular effects between smoked tobacco and cannabis using epinephrine as a measure | Day 2 of each arm
  Urine catecholamine excretion, particularly epinephrine, will be examined in 12-hour urines.
Cardiovascular effects between smoked tobacco and cannabis using platelet activation as a measure | Day 2 of each arm
  We will examine differences in blood and urine biomarkers of platelet activation between smoked tobacco and cannabis.
Cardiovascular effects between smoked tobacco and cannabis using oxidant stress as a measure | Day 2 of each arm
  We will examine differences in blood and urine biomarkers of oxidant stress between smoked tobacco and cannabis.
Cardiovascular effects between smoked tobacco and cannabis using endothelial dysfunction as a measure | Day 2 of each arm
  We will examine differences in blood and urine biomarkers of endothelial dysfunction and inflammation between smoked tobacco and cannabis.
Puffing behaviors across all products | Days 1-2 of each arm
  We will examine how puffing behaviors are different between all products (smoked and vaped cannabis, as well as with smoked tobacco cigarettes) and how they correlate with toxicant biomarker concentrations. Vaping topography measures will be obtained from frame by frame analysis of high definition videos.

CONTACTS AND LOCATIONS:
Overall Officials: Gideon St. Helen, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No